CLINICAL TRIAL: NCT03908957
Title: An Open-label Phase I Clinical Trial to Assess the Safety of Ga68-Dolacga Injection in Healthy Volunteers
Brief Title: to Assess the Safety of Ga68-Dolacga Injection in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Atomic Research Institute, Taiwan (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PTK16081821
Record Dates: First submitted 2019-02-25; First posted 2019-04-09 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Safety Issues

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ga68-Dolacga Injection (Experimental): The healthy volunteer was injected with Ga68-Dolacga Injection iv and performed PET imaging for liver reserve evaluation.
  Interventions: Drug: Ga68-Dolacga Injection

INTERVENTIONS:
Drug: Ga68-Dolacga Injection — Ga68-Dolacga Injection, 3.5±0.25 mCi, single dose iv
  Other Names: Ga68-INER038

SUMMARY:
This is a phase 1 study to evaluate the safety of Ga68-Dolacga Injection in healthy volunteers and to assess the normal reference range and inter-individual variability of the Ga68-Dolacga Injection in estimating liver reserve in healthy volunteers.

DETAILED DESCRIPTION:
Ga-68 is a positron-emitting radionuclide with short half-life of 68 minutes. Dolacga is a non-radiolabeled formulated drug product and will be reconstituted to become the finished radiopharmaceutical product Ga68-Dolacga Injection, a PET tracer specifically targeting to surface receptors of hepatocytes. The study aims to evaluate the safety of Ga68-Dolacga Injection in healthy volunteers and to assess the normal reference range and inter-individual variability of the Ga68-Dolacga Injection in estimating liver reserve in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained before any assessment is performed.
2. Male or female subjects aged 20 or above, inclusive, at date of consent.
3. Body mass index (BMI) between 18.5 and 23.0, inclusive, (BMI will be calculated as weight in kilogram [kg]/height in meters2 [m2])
4. Female subjects must be documented by medical records or physician's note to be either surgically sterile (by means of hysterectomy, bilateral oophorectomy, or tubal ligation) or post-menopausal for at least 1 year or, if they are of child-bearing potential, must commit to use a barrier contraception method for the duration of the study.
5. Male subjects and their partners of childbearing potential must commit to the use of two methods of contraception, one of which is a barrier method for male subjects for the study duration.
6. Male subjects must not donate sperm for the study duration.
7. Willing and able to cooperate with study procedures
8. Physically and mentally healthy subjects as confirmed by an interview, medical history, clinical examination, and ECG
9. Laboratory values within reference range, unless values are deemed by the Principal Investigator as "Not Clinically Significant"
10. Negative result for hepatitis B and C antigen test

Exclusion Criteria:

1. Known or suspected allergy, hypersensitivity, or intolerance to any ingredients of study product as stated in this protocol
2. Implantation of metal devices including cardiac pacemaker, intravascular metal devices
3. Current or prior history of major psychiatric disorders, epilepsy and major depression
4. History of positive test for human immunodeficiency virus (HIV)
5. History of chronic alcohol or drug abuse within the last 6 months
6. Pregnant women, lactating or breast-feeding women
7. Clinically significant abnormal laboratory values and/or clinically significant or unstable medical illness
8. General PET exclusion criteria
9. Prior participation in nuclear medicine treatments or computer tomography examinations in the last year
10. Subject has received an investigational drug or device within 30 days of screening.
11. Subjects having high risks for the study according to the PI discretion
12. Subjects who can't be followed up for any reason

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2019-08-09 (Actual); Study Completion 2019-08-09 (Actual)

PRIMARY OUTCOMES:
Number of subjects reporting clinically significant changes in serum biochemical tests | from pre-dose to 14±2 days post dose
Number of subjects reporting clinically significant changes in hematological tests | from pre-dose to 14±2 days post dose
Number of subjects reporting clinically significant changes in urinalysis | from pre-dose to 14±2 days post dose
Number of subjects with clinically significant changes in systolic blood pressure and diastolic blood pressure | from pre-dose to 14±2 days post dose
Number of subjects with body temperature abnormalities | from pre-dose to 14±2 days post dose
Abnormalities of physical examination in visit 2 (post-treatment) compared with visit 1 | visit 2 (Day 1)
  Including the examination of general appearance, skin, neck (including thyroid), eyes, ears, nose, throat, lungs, heart, abdomen, back, lymph nodes, extremities, vascular and neurological
Number of subjects with clinically significant changes in Heart Rate | from pre-dose to 14±2 days post dose
Number of subjects with clinically significant changes in electrocardiogram(ECG) | from pre-dose to 14±2 days post dose
  The ECG parameters include: PR interval (milliseconds), QTc interval (milliseconds), QRS duration (milliseconds)
Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs) | 14 days
  All laboratory abnormalities which are compared with screening values and out of the reference range will be considered as AE and will be assessed its relationship to the study drug. Any ECG changes including ECG waveform will be assessed as AE(s) and will be followed to assess whether they resolved and when they resolved.

SECONDARY OUTCOMES:
Establishment of the normal reference range of the percent of injection dose (%ID) in healthy liver | up to 60 minutes after administration of Ga68-Dolacga Injection
  The normal reference range will be measured by the mean +/- standard deviation of the liver %ID of all of the phase 1 volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: Yao-Ming Wu, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided